CLINICAL TRIAL: NCT00120874
Title: Memantine and Comprehensive, Individualized, Patient Centered Management of Alzheimer's Disease: A Randomized Controlled Trial
Brief Title: Memantine and Comprehensive, Individualized Management of Alzheimer's Disease and Caregiver Training
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Forest Laboratories (Industry); Fisher Center for Alzheimer's Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H12444-01 A; NAM MD 18 (Other Grant/Funding Number: Forest Laboratories)
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; caregiver training; caregiver counseling; individualized management; memantine; dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Memantine; Exercise; Amyloid beta-Protein Precursor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Individualized Management including caregiver training and Memantine
  Interventions: Behavioral: Individualized management of AD including caregiver training; Drug: Memantine
- Group 2 (Active Comparator): Only Memantine
  Interventions: Drug: Memantine

INTERVENTIONS:
Behavioral: Individualized management of AD including caregiver training — Individualized management program: consists of home visits to get the patient exercising, doing enjoyable activities and cognitive stimulation, educational sessions for caregivers on coping with difficult situations and a caregiver support group to help with questions and emotional concerns.
  Other Names: Namenda; Activity therapy; Cognitive stimulation therapy; Exercise; Caregiver support; Alzheimer's; Alzheimer's Disease
  Arms: Group 1
Drug: Memantine — Patients receive 10 milligrams of memantine twice daily.
  Other Names: Namenda

SUMMARY:
The purpose of this study is to determine whether a comprehensive, individualized management approach with caregiver training and medication with memantine will alleviate symptoms in community dwelling patients with moderate to severe Alzheimer's disease.

DETAILED DESCRIPTION:
Presently some 4.5 million people are afflicted with Alzheimer's disease in the United States. At present pharmacologic treatment, although beneficial, is not curative. Certain nonpharmacologic treatments have assisted caregivers of AD patients by reducing their stress and burden, and others have aided patients, by improving their mood and physical functioning. Comprehensive, individualized approaches to improving Alzheimer's patients' symptomatology and caregiver stress and burden have not been systematically investigated in Alzheimer's patient care. This study seeks to train and counsel caregivers as well as develop an individualized, comprehensive management program that will seek to enhance the functioning of each patient participant.

Patients are randomly placed into one of two groups. Both groups receive memantine and comprehensive evaluations at baseline, 4, 12,28 and 52 weeks. Additionally, group 1 receives an individualized management program, which consists of home visits to get the patient exercising, doing enjoyable activities and cognitive stimulation, educational sessions for caregivers on coping with difficult situations and a caregiver support group to help with questions and emotional concerns.

ELIGIBILITY:
Inclusion Criteria:

* Patients, 50 years of age or greater, residing in the community
* Presence of a family and/or professional caregiver willing and able to participate in all aspects of this study
* A diagnosis of probable Alzheimer's disease by Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) and NINCDS-ADRDA (McKhann,et al., Neurology,1984;34: 939-944) criteria
* A CT or MRI brain scan and medical work up compatible with the DSM-IV and NINCDS-ADRDA diagnostic criteria for Alzheimer's disease
* Mini-Mental State Examination scores of 3-14
* Global Deterioration Scale stages of 5 or 6
* A stage of 6a or greater on the Functional Assessment Staging instrument signifying the presence of dementia deficits in the ability to perform one or more basic activities of daily living

Exclusion Criteria:

* Non-English speaking patients and/or caregivers
* Subjects with a diagnosis of dementia due to conditions other than Alzheimer's disease.
* Subjects with a diagnosis of vascular dementia or a score greater than 4 on the modified Hachinski Ischemic Rating scale
* Patients with a major depressive disorder
* Patients with clinically significant laboratory abnormalities
* Patients receiving investigational pharmacologic agents

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Reisberg, M.D., Principal Investigator — NYU Langone Health; Sunnie Kenowsky, D.V.M., Study Director — NYU Langone Health
Locations (1):
- Fisher Alzheimer's Program, New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Reisberg B, Kenowsky S, Franssen EH, Auer SR, Souren LE. Towards a science of Alzheimer's disease management: a model based upon current knowledge of retrogenesis. Int Psychogeriatr. 1999 Mar;11(1):7-23. doi: 10.1017/s1041610299005554. PMID 10189596
- [Background] Teri L, Gibbons LE, McCurry SM, Logsdon RG, Buchner DM, Barlow WE, Kukull WA, LaCroix AZ, McCormick W, Larson EB. Exercise plus behavioral management in patients with Alzheimer disease: a randomized controlled trial. JAMA. 2003 Oct 15;290(15):2015-22. doi: 10.1001/jama.290.15.2015. PMID 14559955

RESULTS

PARTICIPANT FLOW:
Groups:
- Memantine + CIPCM Program: Individualized Management including caregiver training and Memantine
  Individualized management of AD including caregiver training: Individualized management program: consists of home visits to get the patient exercising, doing enjoyable activities and cognitive stimulation, educational sessions for caregivers on coping with difficult situations and a caregiver support group to help with questions and emotional concerns.
  Memantine: Patients receive 10 milligrams of memantine twice daily.
- Memantine Alone: Only Memantine
  Memantine: Patients receive 10 milligrams of memantine twice daily.
Period: Overall Study
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Started | 10 | 10
Completed Study; Started Extension Study | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Individualized Management and Memantine: Individualized Management including caregiver training and Memantine
  Individualized management of AD including caregiver training: Individualized management program: consists of home visits to get the patient exercising, doing enjoyable activities and cognitive stimulation, educational sessions for caregivers on coping with difficult situations and a caregiver support group to help with questions and emotional concerns.
  Memantine: Patients receive 10 milligrams of memantine twice daily.
- Memantine: Only Memantine
  Memantine: Patients receive 10 milligrams of memantine twice daily.
- Total: Total of all reporting groups
Arm/Group | Individualized Management and Memantine | Memantine | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 9 | 10 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic-American | 0 | 2 | 2
  White, not of Hispanic-American Origin | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinician Interview-Based Assessment of Change Plus Caregiver Input (CIBIC-Plus) Global Score (New York Univeristy Version)
Description: CIBIC-Plus is measured in units on a scale ranging from 1 to 7, where 1 is markedly improved, 4 is unchanged, and 7 is markedly worse
Time Frame: Baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 2.3 (1.16) | 5.22 (1.56)

2. Primary Outcome: Change From Baseline in Clinician Interview-Based Assessment of Change Plus Caregiver Input (CIBIC-Plus) Global Score (New York Univeristy Version)
Description: as for outcome 1
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 2.1 (1.45) | 6 (1.32)

3. Secondary Outcome: Change From Baseline of the Severe Impairment Battery (SIB)
Description: The SIB evaluates cognitive performance. It is a 51 item scale which assesses social interaction, memory, language, orientation, attention, praxis, visuospacial ability and construction. Scores range from 0 (greatest impairment) to 100 (least impairment).
Time Frame: Baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 51.3 (33.843) | 54 (37.002)

4. Secondary Outcome: Change From Baseline of the Severe Impairment Battery (SIB)
Description: as for outcome 3
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 45.1 (33.365) | 48 (37.353)

5. Secondary Outcome: Change From Baseline of the Mini-Mental State Examination (MMSE)
Description: The MMSE is a graded on a 30 point scale that measures cognitive functioning. A lower score indicates a higher level of impairment. Complete scale range is -no cognitive impairment=24-30; mild cognitive impairment=18-23; severe cognitive impairment=0-17.
Time Frame: Baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 6.7 (5.143) | 8.4 (5.816)

6. Secondary Outcome: Change From Baseline of the Mini-Mental State Examination (MMSE)
Description: as for outcome 5
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 6.7 (4.138) | 6.7 (5.477)

7. Secondary Outcome: Change From Baseline of the Functional Assessment Staging Disability Score (FAST-DS)
Description: The FAST-DS assesses the magnitude of progressive functional deterioration by identifying characteristic progressive disabilities in participants with AD. Scores range from 1.0 (normal) to 7f (severe loss of ability, not even able to hold up head independently). Scores are made up of stages (1 through 7) and substages (from a to e for stage 6; from a to f for stage 7). The following scoring for substages is applied: 6a=6.0, 6b=6.2, 6c=6.4, 6d=6.6, 6e=6.8, 7a=7.0, 7b=7.2, 7c=7.4, 7d=7.6, 7e=7.8, 7f=8.0. Additionally, non-consecutive deficits are noted and scored as follows: full stage non-consecutive deficit=1.0, non-consecutive substage deficit=0.2.
  The overall FAST-DS score = (FAST Stage Score) + (Each Non-Consecutive FAST disability scored as described)
Time Frame: Baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 6.16 (0.631) | 6.67 (0.246)

8. Primary Outcome: Change From Baseline of The Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory Modified for Severe Dementia Abbreviated Version (ADCS-ADLsev-abv)
Description: The ADCS-ADLsev-abv is a structured questionnaire where each item consists of a series of hierarchical questions designed to determine a patient's ability to perform the activities of daily living as assessed by the caregiver. Possible scores range from 0 to 39, where a higher score is indicative of greater capacities.
Time Frame: Baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 21.9 (8.034) | 9.6 (6.041)

9. Primary Outcome: Change From Baseline of The Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory Modified for Severe Dementia Abbreviated Version (ADCS-ADLsev-abv)
Description: as for outcome 8
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 18.5 (8.045) | 7.6 (6.766)

10. Secondary Outcome: Change From Baseline of the Functional Assessment Staging Disability Score (FAST-DS)
Description: as for outcome 7
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 6.5 (0.254) | 6.84 (0.279)

11. Secondary Outcome: Change From Baseline of The Behavioral Pathology in Alzheimer's Disease Frequency Weighted Severity Scale (BEHAVE-AD-FW)
Description: The BEHAVE-AD-FW measures the frequency and severity of 25 behavioral symptoms with a total score and global rating. Individual behavioral assessments are rated for severity (0=none to 3-most severe) and frequency (1=least frequent to 4=most frequent) which are then multiplied; scores for each of the 25 items are then summed. Possible total scores range from 0 to 297. The global rating is scored from 0 (not dangerous to patient, not troubling to caregiver) to 3 (dangerous to patient, highly troubling to caregiver). Global rating was not analyzed for this study. The higher the score the worse the outcome.
Time Frame: Baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 7.2 (5.308) | 23.7 (14.952)

12. Secondary Outcome: Change From Baseline of The Behavioral Pathology in Alzheimer's Disease Frequency Weighted Severity Scale (BEHAVE-AD-FW)
Description: The BEHAVE-AD-FW measures the frequency and severity of 25 behavioral symptoms with a total score and global rating. Individual behavioral assessments are rated for severity (0=none to 3-most severe) and frequency (1=least frequent to 4=most frequent) which are then multiplied; scores for each of the 25 items are then summed. Possible total scores range from 0 to 297. The global rating is scored from 0 (not dangerous to patient, not troubling to caregiver) to 3 (dangerous to patient, highly troubling to caregiver). The higher the score the worse the outcome.
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 8.1 (5.131) | 21.2 (11.893)

13. Secondary Outcome: Change From Baseline of the Revised Memory and Behavior Problems Checklist (RMBPC): Frequency
Description: The RMBPC is a 24 item rating scale of the frequency of memory and behavioral problems in the AD subject and of how upset or "bothered" their caregivers react. Frequency is rated from 0 (least frequent) to 4 (most frequent) and caregiver reaction is rated from 0 (not at all) to 4 (extremely bothered or upset). Higher scores indicate more frequent memory and behavioral problems in the subject with AD as well as a more upset or bothered caregiver. Possible scores range from 0 to 96.
Time Frame: Baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 24.7 (9.945) | 34.9 (9.515)

14. Secondary Outcome: Change From Baseline of the Revised Memory and Behavior Problems Checklist (RMBPC): Caregiver Reaction
Description: as for outcome 13
Time Frame: Baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 2.0 (2.582) | 10.7 (14.143)

15. Secondary Outcome: Change From Baseline of the Revised Memory and Behavior Problems Checklist (RMBPC): Frequency
Description: as for outcome 13
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 24.4 (8.449) | 32.4 (11.4)

16. Secondary Outcome: Change From Baseline of the Revised Memory and Behavior Problems Checklist (RMBPC): Caregiver Reaction
Description: as for outcome 13
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine + CIPCM Program | Memantine Alone
Number analyzed (Participants) | 10 | 9
units on a scale | 3.8 (6.68) | 11.4 (11.599)

ADVERSE EVENTS:
Arm/Group | Individualized Management and Memantine | Memantine
Serious Adverse Events (participants affected / at risk) | 3/10 | 10/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individualized Management and Memantine (N=10) | Memantine (N=10)
Left Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Infections and infestations) | 0 (0) | 1 (1) — C. dificil infection
Left heel Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Left heel Infection (Infections and infestations) | 0 (0) | 1 (1)
Left Pelvic Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stage II Pressure Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Located above Anus to tail bone
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospitalized, determined by CT scan
Urinary tract Infection (Infections and infestations) | 0 (0) | 1 (1) — No growth on Culture and sensitivity
Dehydration (General disorders) | 0 (0) | 1 (1)
Cardiopulmonary Arrest (General disorders) | 0 (0) | 1 (1) — Unexpected event
Atherosclerotic Heart Disease (General disorders) | 0 (0) | 1 (1) — Vascular disorders Cardiac disorders
Syncope (General disorders) | 0 (0) | 2 (4) — 1 Subject had 2 episodes & was placed in hospice. 2nd subject had 2 syncopal episodes, 1 at a restaurant & 2nd episode in Dr. office
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individualized Management and Memantine (N=10) | Memantine (N=10)
abnormal blood results (Investigations) | 1 (1) | 0 (0) — slightly low copper, low zinc, mild elevation of serotonin
red blotch on face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — lasted 2-3 hours
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) — Treated with antibiotics
Dizziness (General disorders) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Diarrhea (Infections and infestations) | 1 (1) | 1 (2) — C. dificil
Fungal skin rash in groin (Infections and infestations) | 1 (1) | 0 (0)
toenail fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Calcified bone mass on hip due to muscle tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
abnormal urine analysis (Investigations) | 1 (1) | 0 (0) — possible urinary tract infection
Vitamin D insufficiency (General disorders) | 1 (1) | 0 (0)
Rigidity (Nervous system disorders) | 0 (0) | 2 (2) — 1 subject had Parkinsonian symptoms of rigidity and instability, a second subject had rigidity possibly due to supplement usage
Abnormal sensation in hands (Nervous system disorders) | 0 (0) | 1 (1)
Increasing hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) — Subject was euthyroid at baseline on medication & later diagnosed with hypothyroidism
Increased alkaline phosphatase (Investigations) | 0 (0) | 2 (3) — 1 subject had an increased alkaline phosphatase at 2 study visits, a second subject had an elevated alkaline phosphatase at 1 visit
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (5) — 3 subjects each had 1 episode of constipation reported by caregiver, a 4th subject had 1 episode determined by hosp dr, a 5th subject had chronic constipation reported once,
Elevated Platelet Count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Black blister on Left heel (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 4 (4) — 4 subjects were reported to have difficulty swallowing pills.
Brown liquid coming from nose (General disorders) | 0 (0) | 1 (1) — Occurred simultaneously with diarrhea
Sleepiness (General disorders) | 0 (0) | 1 (1)
Decreased appetite (General disorders) | 0 (0) | 1 (2) — 1 subject had dec appetite in general once starting carbidopa/levodopa, a 2nd subject stopped eating for 2 days then had a decreased appetite afterwards
Electrolyte abnormality (General disorders) | 0 (0) | 1 (1) — elevated calcium
Hearing Loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) — 1 subject developed hearing loss when started taking Namenda
Increased leg edema (General disorders) | 0 (0) | 1 (1) — 1 subject had mild leg edema at baseline and it was reported to have worsened at Wk 4 study visit
Cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) — 1 subject had 1 episode,a 2nd subject had 2 episodes,
Stage I Pressure Sore (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (2) — 1 subject had 2 episodes which occurred concurrently with syncope and hypotension
Hypotension (General disorders) | 0 (0) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 1 (1) — 1 subject fell out of bed
Bruised ribs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — 1 subject from falling out of bed. Dx on PE by Dr.
Buttocks abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Buttocks ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Elevated creatinine and decreased GFR (Investigations) | 0 (0) | 1 (1)
Hypoglycemia (General disorders) | 0 (0) | 2 (2) — 1 subject had 1 asymptomatic episode on Wk 4 bloodwork, 1 subject had mild hypoglycemia
Elevated C Reactive Protein (General disorders) | 0 (0) | 1 (1) — Cause not found
mild hypercholesterolemia (Investigations) | 0 (0) | 1 (1)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — CT scan
Adipsia (General disorders) | 0 (0) | 1 (1) — Lasted 2 days
Lost ability to walk (General disorders) | 0 (0) | 1 (1) — Occurred simultaneously with syncopal event
Lip smacking and chomping (General disorders) | 0 (0) | 1 (2) — Occurred continuously, reported at 2 study visits wk4 & wk12
Skin tear (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — RLE
Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Right hip

LIMITATIONS AND CAVEATS:
The original statistician who worked on this study left the institution prior to completing data analysis. A new statistician has been engaged. In the unlikely event that outcome measures data changes, it will be updated accordingly in this record.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes